CLINICAL TRIAL: NCT04773535
Title: Validation of the DyCare® Lynx System for Motion Analysis of the Wrist During Standard Movements and Daily Activities
Brief Title: Validation of the DyCare® Lynx System for Motion Analysis of the Wrist
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2018-00457
Record Dates: First submitted 2020-11-19; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy Volunteers: Adult (>18y) healthy volunteers without previous injuries or pathologies of the hand and upper extremity
  Interventions: Device: 3D Motion analysis

INTERVENTIONS:
Device: 3D Motion analysis — Motion analysis using DyCare® Lynx system with inertial based sensors as well as an optoelectronic motion analysis system based on infrared cameras (11x Vicon infrared high speed cameras)

SUMMARY:
This project is set to compare the wrist joint movement measurements of the DyCare® Lynx System with optoelectronic motion analysis using a marker system and infrared cameras.

A total of 10 healthy test persons will be subjected to both the DyCare® Lynx and the Vicon® measurements during standard movements as well as during activities of daily living. The wrist joint angles measured with both systems will be compared.

DETAILED DESCRIPTION:
The accepted laboratory gold standards for human motion analysis are too over-elaborated for clinical use. The DyCare® Lynx system is user-friendly and has been proven reliable for motion evaluation of different joints, but not yet for the wrist.

Therefore, this project is set to compare the wrist joint movement measurements of the DyCare® Lynx System with optoelectronic motion analysis using a marker system and infrared cameras. DyCare® Lynx is based on two inertial sensors (DyTrack) capable of objectively measuring three dimensional joint movements in real time. Each inertial sensor includes an accelerometer, gyroscope and magnetometer and captures up to 1'000 samples per second. DyCare® Lynx is certified for measurements on the human musculoskeletal apparatus (EN ISO 13485:2003 Certificate No. 15185 - M), is CE marked and will only be applied to each participant for a few minutes during the measurements. The control measurements will be conducted using a Vicon® motion capture system in the Motion Analysis Laboratory of the Department of Plastic Surgery and Hand Surgery of the University Hospital of Zurich. The Vicon® system is equipped with 11 infrared cameras. The system is made for 'Life science application' and is approved as CE medical device. A total of 10 healthy test persons will be subjected to both the DyCare® Lynx and the Vicon® measurements during standard movements as well as during activities of daily living. The wrist joint angles measured with both systems will be compared, therefore limits of agreement, maximum difference and root mean squared difference will be calculated to quantify the deviation between methods. The standard error of measurements will be calculated to determine repeatability of the systems.

ELIGIBILITY:
Inclusion Criteria:

* 10 test persons with healthy right-dominant hands
* Test Persons older than 18 Years
* Test persons willing and able to give written informed consent to participate in the study

Exclusion Criteria:

* Inflammatory disease (e.g. rheumatoid arthritis)
* German language barrier to understand instructions
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Legal incompetence
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Active wrist movement at standard movements | October 2019
  Ten healthy subjects will be recorded (3D motion analysis) while performing flexion-extension and radial-ulnar deviation movements of their right wrist using inertial sensors and skin markers

SECONDARY OUTCOMES:
Active Wrist movement during activities of daily living. | January 2020-August 2021
  Ten healthy subjects will be recorded (3D motion analysis) while performing during ADLs: opening a jar, opening a lid pot, turning a key, dart-throwing.
Comfort of the wearable Sensors | October 2019
  questionnaire looking into six dimensions of comfort as proposed by Knight and Baber (Knight, J.F.; Baber, C. A tool to assess the comfort of wearable computers. Human Factors 2005, 47, 77-91, doi:10.1518/0018720053653875.
Time Consumption of measurements using DyCare® Lynx | October 2019
  Minutes necessary to attach the sensors to the patients and to record the movements.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, PD Dr. med, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Clinic of Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided